CLINICAL TRIAL: NCT06914258
Title: Effects of Inhibition Compression Versus Scapular Mobilization Technique on Shoulder in Patients With Mastectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/818
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Mastectomy; Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhibition Compression (Experimental)
  Interventions: Combination Product: Inhibition Compression
- Scapular Mobilization Technique (Experimental)
  Interventions: Combination Product: Scapular Mobilization Technique

INTERVENTIONS:
Combination Product: Inhibition Compression — Group A will receive conventional Physiotherapy treatment along with the scapular mobilization which will include;
  * Electrotherapy (TENS and hot pack) for 10 min
  * Active and passive ROMs for 5 min
  * pectoral stretching for 5min
  * shoulder joint mobilization. To mobilize the shoulder joint, distraction of the glenohumeral joint, posterior glide and caudal glide were performed to the patient in supine position at a frequency of two to three oscillations/second for one to two minutes. (10 min)
  * Manual scapular mobilization will be done in sideline with their back towards the physiotherapist.
  Arms: Inhibition Compression
Combination Product: Scapular Mobilization Technique — Group B will receive the same baseline physiotherapy treatment as in group A along with the Inhibition compression therapy which is a (MET). MET was performed on shoulder. Patient position: supine lying position. Following are the steps involved in application of MET: (1) stretch the muscle to a felt 'barrier' or to their tolerance of stretching (2) create a voluntary contraction that is isometric of the muscle being stretched while being resisted with equal and regulated counterforce by the physiotherapist for 7-10 seconds. (3) a stretch is held for a set amount of time after the muscle relaxes (4) the physiotherapist "takes up the slack" once the muscle relaxes Duration of treatment was approximately 15-20 minutes.
  Arms: Scapular Mobilization Technique

SUMMARY:
A mastectomy is a medical surgery in which the breast is removed whole or in part. Breast cancer is the second most prevalent cancer diagnosed in women. Rotator cuff dysfunction-related shoulder pain is a common symptom associated with mastectomy, reconstruction, and therapy for breast cancer.) Patients who get treatment for breast cancer report reduced strength (prevalence 17-33%), loss of upper limb range of motion (prevalence 2-51%), and reduced ability to carry out daily life tasks.

DETAILED DESCRIPTION:
The study aims to observe the effectiveness of inhibition compression therapy versus scapular mobilization on shoulder in patients with mastectomy. By investigating the effectiveness of inhibition compression therapy versus scapular mobilization, this study can contribute to improved pain management, enhanced quality of life, and reduced healthcare utilization for breast cancer survivors. It will be randomized control trial (RCT). The study will be conduct in Gujranwala institute of nuclear medicine. It will be non-probability convenience sampling technique. Duration of the study will be 6 months after the approval of synopsis

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 75 years (42)
* unilateral breast cancer followed by chemotherapy or radiations. (27)
* modified radical mastectomy surgery (27)
* limited ROM of shoulder
* Female

Exclusion Criteria:

* Patients with recurrent breast cancer (42)
* History of ischemic heart disease
* History of high blood pressure
* History of other surgery
* Any neurological issue

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 12 Months
  Patients complete the 13-item Shoulder discomfort and Disability Index (SPADI) to gauge their level of discomfort and degree of difficulty doing activities of daily living (ADLs) that require the use of their upper extremities. There are five items on the pain subscale and eight items on the disability subscale. The following patient demographics can benefit from SPADI use: pain in the shoulders Rotator cuff injury, Osteoarthritis, rheumatoid arthritis, Shoulder Frozen and Shoulder replacement.
  Using the affected shoulder, the patient is asked to select the number that most accurately represents their degree of pain and difficulty. The sum of the disability and pain scales is 80 and 50, respectively. The percentage represents the overall SPADI score.
  A score of 100 denotes the worst, while 0 denotes the finest. A higher score indicates greater disability
Constant-Murley Shoulder Outcome Score | 12 Months
  The Constant-Murley score (CMS) is a scale of 100 points made up of several distinct characteristics. These factors determine the patient's degree of pain and capacity to perform everyday tasks. To assess functionality following shoulder injury treatment, the Constant-Murley score was developed. The test is broken down into four subscales: range of motion (forward elevation, external rotation, abduction, and internal rotation of the shoulder) (40 points), activities of daily life (20 points), and discomfort (15 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Gujranwala institute of nuclear medicine, Gujranwala, Pakistan

IPD SHARING:
Plan to Share IPD: No